CLINICAL TRIAL: NCT02268370
Title: Treatment-free Remission Accomplished With Dasatinib in Patients With CML
Acronym: TRAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ozmosis Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BMS CA180-543; OZM-056 (Other: Ozmosis Research Inc.)
Record Dates: First submitted 2014-09-25; First posted 2014-10-20 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Other): This research is being done because dasatinib has been shown to achieve a deep molecular response in patients as compared to imatinib.
  Patients in this study will continue to take their own supply of imatinib for three months to ensure they have achieved a stable response to the drug. Once this has been confirmed, imatinib will be stopped and the patients in this study will then be monitored to see if their CML relapses. This period can last up to 2.5 years.
  If the participant has a relapse, they will be started on dasatinib and will continue to receive dasatinib for up to 2 years.
  If after one year they achieve a response, they will continue on dasatinib for one more year. If the participant maintains this response, they will have the option of discontinuing dasatinib.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib
  Other Names: Sprycel

SUMMARY:
The purpose of this study is to find out how to increase the potential for achieving an "operational cure" from chronic myeloid leukemia. An "operational cure" is a state in which a person does not require further treatment, although there may be some remaining cancer cells. Patients would normally remain on a TK inhibitor indefinitely within a standard of care setting for chronic myeloid leukemia. Within this clinical trial, patients will discontinue their TK inhibitor prematurely. If any signs of progression are identified, dasatinib will be introduced.

This research is being done because dasatinib has been shown to achieve a greater response in a much higher proportion of patients as compared to imatinib. Dasatinib is approximately 300 times more potent than imatinib, and it is possible that a greater response can be achieved by dasatinib than by imatinib.

DETAILED DESCRIPTION:
This is an open label, single arm Phase II trial that will examine how safe and effective it will be for patients with chronic myeloid leukemia (CML) to discontinued first line tyrosine kinase inhibitor (TKI) therapy.

The main goal of this study is to determine the potential role of dasatinib (the study drug) in helping patients with CML attain a sustained treatment free remission.

During this study the safety and tolerability of Dasatinib will be evaluated by means of drug related toxicity, adverse event reports, physical examinations and laboratory safety evaluations.

The study period for an individual patient is expected to be approximately between 30-72 months.

A total of 135 patients will be recruited from 10 Canadian centres.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CML
2. Treatment of chronic phase CML treated for a minimum of three years exclusively with imatinib
3. Levels of BCR-ABL by RQ-PCR with ≥ 4.5 log reduction from baseline
4. Provide written informed consent
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
6. Age >18 years.
7. Adequate organ liver and renal functions
8. Normal serum levels (within normal limits)

Exclusion Criteria:

1. Prior treatment with a TKI (except for imatinib, hydroxyurea, anagrelide or interferon)
2. Taking any medications or substances known to affect CYP3A4.
3. Concurrent medical condition which may increase the risk of toxicity
4. History of significant bleeding disorder unrelated to cancer
5. Cardiac Symptoms
6. Clinically significant hypokalemia or hypomagnesemia that cannot be corrected prior to dasatinib administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2014-10; Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Molecular Remission | change from baseline in Molecular Profile at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kim, MD, Principal Investigator — University Health Network, Toronto
Locations (12):
- Canada (12):
  - Tom Baker Cancer Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hôpitallier Universitaire de Quebec - Hôpital de l'Enfant-Jésus, Charlesbourg, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec